CLINICAL TRIAL: NCT04228510
Title: The Role of Two- Dimensional Speckle Tracking Echocardiography in Prediction of Remodeling and Major Adverse Cardiovascular Events in ST Elevation Myocardial Infarction After Primary Percutaneous Coronary Intervention
Brief Title: Two- Dimensional Speckle Tracking Echocardiography After Primary Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Rafat Rasmy, Principal investigator, Assiut University
Other Study IDs: 2DSE
Record Dates: First submitted 2020-01-12; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: ST elevation myocardial infarction (STEMI) patients after primary percutaneous coronary intervention who will be followed up in Assiut University hospital.
  Interventions: Procedure: 2D speckle tracking echocardiography

INTERVENTIONS:
Procedure: 2D speckle tracking echocardiography — Global and segmental strain and strain rate in longitudinal and circumferential directions will be detected after PPCI; before discharge. The LV circumferential strains and strain rates will be determined from the short-axis views at the basal, middle, and apical levels, and longitudinal strains and strain rates will be determined from the apical 2-, 3-, and 4-chamber views of the LV.
  Segmental longitudinal strains equal to -15% or closer to 0 will be considered abnormal (injured segments). The average segmental longitudinal strain and strain rate of the abnormal segments is defined as the injury longitudinal strain (InjLS) and injury longitudinal systolic strain rate (InjLSRs).

SUMMARY:
ST-segment elevation myocardial infarction (STEMI) is a major cause of morbidity and mortality worldwide. In spite of decrease in acute and long-term mortality following STEMI in parallel with more use of reperfusion therapy, such as primary percutaneous coronary intervention (PPCI), modern antithrombotic therapy, and secondary prevention, mortality remains considerable. Reduced EF is a well-known predictor of increased short and long term major adverse cardiovascular events MACE :( heart failure, stroke and death)

ELIGIBILITY:
Inclusion Criteria:

* ST elevation myocardial infarction patients after primary percutaneous coronary intervention

Exclusion Criteria:

* Previous myocardial infarction.
* Sever or haemodynamically significant (associated with chamber dilation) valvular heart diseases.
* Previous heart failure.
* Previous cerebrovascular strokes.
* Atrial fibrillation.
* Severe comorbidities as severe renal impairment, hepatic or respiratory failure.
* Bad equality views which affects accurate speckle tracking imaging.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ST elevation myocardial infarction patients after primary percutaneous coronary intervention who will be followed up for a one year in Assiut University hospital.
Sampling Method: Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The Incidence of major adverse cardiovascular events | 1 year
  the rate of Acute coronary syndrome, Heart failure, Stroke and all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Helmy, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No